CLINICAL TRIAL: NCT01083511
Title: Collection & Extraction of Respiratory Specimens for the Validation of the Artus Influenza RG PCR Test
Brief Title: Collection and Extraction of Respiratory Specimens
Status: Completed | Type: Observational
Sponsor: QIAGEN Gaithersburg, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: C09-INFLUENZA-002
Record Dates: First submitted 2010-03-08; First posted 2010-03-09 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Influenza
Keywords: Influenza; Influenza A; Influenza B; Swine Influenza A/H1N1; Respiratory Virus
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Extracted nucleic acid, Residual Universal Transport Medium.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Symptomatic: Individuals with signs and symptoms of a respiratory tract infection where it is suspected that such signs and symptoms are caused by a respiratory virus infection.

SUMMARY:
The study will be conducted with nasopharyngeal swab specimens collected prospectively from individuals suspected of having an acute respiratory tract infection caused by an Influenza virus. A series of standard viral culture tests validated for routine use in the clinical laboratory, as well as the CDC swine H1N1 test will be used to establish a collection of well characterized specimens. For each specimen four (4) aliquots will be prepared. One aliquot will be tested in real-time using the requisite viral culture reference methods, one aliquot will be used for H1N1 reference testing, one aliquot will be used to extract nucleic acid in real-time, and one aliquot of the UTM will be archived for the purpose of sequencing to confirm Influenza-positive specimens. The extracted nucleic acid and any remaining specimen will be stored at -70°C for later testing by the artus Influenza RG PCR test, or other investigational method(s).

DETAILED DESCRIPTION:
Each year the morbidity and mortality associated with respiratory tract infections fluctuates seasonally. This rise and fall is associated with the changing prevalence of respiratory viruses in the population. Myriad respiratory viruses are responsible for these infections. For example, Influenza Virus, Respiratory Syncytial Virus (RSV), Parainfluenza Virus, Human Metapneumovirus, Rhinovirus, and Adenovirus have all been identified as causing such infections. Numerous pathogenic subtypes have been identified within most of these viral groups. Apart from supportive measure (e.g., bed rest, hydration, etc.), there are no effective treatments for these viral infections; however, antiviral agents (e.g.,Tamiflu) can be used to alleviate the severity of flu-like symptoms.

Each year the virus population fluctuates, and with it the antigenic presentation of the dominant strains that circulate through the population. Epidemics arise when larger and larger portions of the population do not have innate or acquired resistance to such strain(s) in a given season. The World Health Organization (WHO) maintains a separate website dedicated to tracking outbreaks of influenza, especially avian influenza (https://www.who.int/fluvirus_tracker). Influenza outbreaks monitored in the hope that a pandemic similar to the Spanish Flu of 1918 can be avoided; it is estimated that well over 25 million people died from the Spanish Flu. The United States government also maintains a separate website with resources regarding the flu and pandemic related information (http://www.pandemicflu.gov/). On June 11, 2009 the WHO raised the pandemic threat level to 6 in response to the global appearance of a new strain of swine Influenza A (subtype H1N1). The rapidity with which the H1N1 virus has spread exemplifies the notion that quickly and accurately identifying a viruses associated with an outbreak is critical to global public health.

In the present study a collection of respiratory specimens that are well characterized will be archived for later evaluation using the artus® Influenza RG PCR test. The artus Influenza test is a real-time PCR test that identifies Influenza A, Influenza B, and Influenza Type A/subtype H1N1 from nasopharyngeal swab specimens.

ELIGIBILITY:
Inclusion Criteria:

* Subjects that sign the Informed Consent form required for prospectively enrolling patients into the study.
* Subjects that present at a hospital, clinic, or physician's office with symptoms of a respiratory tract infection.
* Subjects with an acute respiratory infection where said acute respiratory infection is suspected of being caused by an Influenza virus.

Exclusion Criteria:

- Subjects where the duration of the symptoms of such an acute respiratory infection is greater than or equal to 7 days (i.e., ≥7).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes individuals having the signs and symptoms of a respiratory tract infection caused by an Influenza virus.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2010-03; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Presence of Influenza Virus | Specimens will be taken within 7 days of the appearance of symptoms.
  To confirm the presence of Influenza virus in nasopharyngeal specimens taken from individuals having influenza like symptoms.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Arizona, Tucson, Arizona
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Ohio State University, Columbus, Ohio